CLINICAL TRIAL: NCT04633070
Title: Use of Gamification in Health Apps for Lifestyle Intervention: A Systematic Review
Brief Title: Systematic Review of Health App Gamification for Lifestyle Intervention Adherence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CCS-Health Apps 2020
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Mobile Applications; Diet, Healthy; Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Gamification — Gamification (including, but not limited to a ranking system, badges and achievements, points, social media interaction, and leveling up) within mobile and web-based applications (also referred to as 'apps') for lifestyle modification (diet, physical activity, smoking cessation etc).

SUMMARY:
Health behaviour applications (also referred to as "apps") have the potential to provide several advantages for motivating behaviour change for health and well-being. Finding ways to increase and sustain health promoting behaviour changes has been a challenge during health app development. Gamification, which is the use of game elements in a non-game situation, shows promise and has proven effective in many fields. However, key questions remain concerning how to use gamification in apps to modify health behaviour, especially to support adherence to dietary pattern recommendations. To investigate and summarize the current evidence, a systematic review of the totality of evidence from clinical trials and observational studies will be conducted to capture and distinguish the types of gamification strategies that may be most effective in improving and sustaining health promoting behaviours to inform future health behaviour app development.

DETAILED DESCRIPTION:
Background: Studies on health behaviours such as physical activity and smoking cessation (behaviour change) have indicated that gamification is an effective tool for engagement and behaviour change, especially when multiple different competitive elements are used including: a ranking system, badges and achievements, points, social media interaction, and leveling up. Gamification is the use of game elements in a non-game environment to invoke behaviour change. The majority of health-focused gamification investigations are currently conducted using web or mobile-based delivery platforms in adults focusing on physical activity. Access to these web and mobile based applications through smartphones, tablets and computers has grown rapidly. In 2016, 94% of Canadians had home internet access, with 88% reporting that they use a smartphone for personal use. Moreover, a recent survey in the US found that 73% of those with, or at risk of cardiovascular disease, have a smartphone and 43% use a health-related application to track progress towards a health goal. While research on mobile-based app use for modifying diet is promising, the effectiveness of using gamification in apps for sustaining dietary pattern adherence is unclear. An investigation and summary of the current types of gamification strategies that may be most effective is important to inform and aid future app development. The ultimate aim of this research investigation is to inform the development of the PortfolioDiet.app, a dietary pattern adherence application for reducing LDL-cholesterol in individuals at risk for cardiovascular disease.

Objective: To conduct a systematic review investigating the gamification strategies used in applications for long term behaviour change, with a specific focus on dietary pattern adherence in adults.

Design: A systematic review of the literature will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: The investigators will include prospective cohort studies and controlled trials. Studies will be included if they are >= 2-months in duration and assess the relation of different gamification strategies used in health behaviour applications with adherence to the health intervention, participant engagement with using the application, and/or the intended health outcome. There will be no language restrictions.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus.

Outcomes: The primary outcome will be adherence to the intervention associated with use of the application, such as, but not limited to: physical activity, smoking cessation, increasing fruit and vegetable intake, improving healthy food index score. Secondary outcomes will include participant engagement with use of the application. This adherence to using the application may be determined based on number of using days using the application compared to intended number of days of application usage. Observation of a significant change in the intended health outcome, such as, blood glucose, HbA1c, blood lipids, weight change [BMI, body weight, waist circumference, will also be assessed.

Data Synthesis: A Microsoft Excel spreadsheet will be used to track the extractions and summarize the qualitative and quantitative data from each study.

Risk of Bias (Quality) Assessment: The risk of bias of each included study will be assessed using the Cochrane Handbook for Systematic Reviews of Interventions. This will be done in relation to evaluating the criteria for assessing risk as either low, high or uncertain risk of bias as identified in the Risk of Bias tool.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national and international scientific meetings and publication. As well as utilized in a publically available web-based application hosted on the Canadian Cardiovascular Society website.

Significance: Gamification has been identified as a promising tool for health promotion. While research directly comparing gamified interventions to non-gamified controls has found beneficial effects on physical activity, or more recently mental health, there is a lack of evidence on investigating gamification for dietary change. As poor health behaviours (i.e. unhealthy diet, smoking, sedentary behaviour) have been repeatedly identified as major contributors to disease burden in Canada and globally, interventions which can target and improve these behaviours over a long term are required. Furthermore, as the generations who have grown up with the internet and app technology begin to age they will seek engaging digital tools to improve health outcomes, and therefore the need for digital health interventions that are effective at improving and sustaining beneficial health behaviours will only continue to grow.

ELIGIBILITY:
Inclusion Criteria for controlled trials:

* Randomized and non-randomized controlled intervention studies in humans
* Gamification intervention
* Presence of an adequate comparator, such as standard of care or an application without gamification components
* Intervention duration >=2 months
* Viable outcome data

Inclusion Criteria for prospective cohort studies:

* Prospective cohort studies
* Duration >= 2-months
* Assessment of the exposure of gamification used in a health behaviour application
* Ascertainment of viable outcome data by level of exposure

Exclusion Criteria for controlled trials:

* Lack of an adequate comparator
* Non-health behaviour application

Exclusion Criteria for prospective cohort studies:

* Ecological, cross-sectional, or retrospective observational studies
* Intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults (>=18 years), regardless of health status.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Adherence to the intervention | At least 2 months
  Percentage change

SECONDARY OUTCOMES:
Participant app engagement | At least 2 months
  Adherence to using the app based on number of using days using the app compared to intended number of days of app usage
Health outcome - body weight | At least 2 months
  Weight change
Health outcome - BMI | At least 2 months
  BMI change
Health outcome - body fat | At least 2 months
  Body fat change
Health outcome - waist circumference | At least 2 months
  Waist circumference
Health outcome - HbA1c | At least 2 months
  HbA1c change
Health outcome - fasting plasma glucose (FPG) | At least 2 months
  FPG change
Health outcome - LDL-cholesterol (LDL-C) | At least 2 months
  LDL-C change
Health outcome - non-HDL-cholesterol (non-HDL-C) | At least 2 months
  Non-HDL-C change
Health outcome - apoB | At least 2 months
  ApoB change
Health outcome - HDL-cholesterol (HDL-C) | At least 2 months
  HDL-C change
Health outcome - triglycerides | At least 2 months
  Triglycerides change
Health outcome - systolic blood pressure (SBP) | At least 2 months
  SBP change
Health outcome - diastolic blood pressure (DBP) | At least 2 months
  DBP change

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam S, Lang JJ, Drucker AM, Gotay C, Kozloff N, Mate K, Patten SB, Orpana HM, Afshin A, Cahill LE. Assessment of the burden of diseases and injuries attributable to risk factors in Canada from 1990 to 2016: an analysis of the Global Burden of Disease Study. CMAJ Open. 2019 Feb 28;7(1):E140-E148. doi: 10.9778/cmajo.20180137. Print 2019 Jan-Mar. PMID 30819694
- [Background] El-Hilly AA, Iqbal SS, Ahmed M, Sherwani Y, Muntasir M, Siddiqui S, Al-Fagih Z, Usmani O, Eisingerich AB. Game On? Smoking Cessation Through the Gamification of mHealth: A Longitudinal Qualitative Study. JMIR Serious Games. 2016 Oct 24;4(2):e18. doi: 10.2196/games.5678. PMID 27777216
- [Background] GBD 2017 Risk Factor Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1923-1994. doi: 10.1016/S0140-6736(18)32225-6. Epub 2018 Nov 8. PMID 30496105
- [Background] Johnson D, Deterding S, Kuhn KA, Staneva A, Stoyanov S, Hides L. Gamification for health and wellbeing: A systematic review of the literature. Internet Interv. 2016 Nov 2;6:89-106. doi: 10.1016/j.invent.2016.10.002. eCollection 2016 Nov. PMID 30135818
- [Background] Cumpston M, Li T, Page MJ, Chandler J, Welch VA, Higgins JP, Thomas J. Updated guidance for trusted systematic reviews: a new edition of the Cochrane Handbook for Systematic Reviews of Interventions. Cochrane Database Syst Rev. 2019 Oct 3;10(10):ED000142. doi: 10.1002/14651858.ED000142. No abstract available. PMID 31643080
- [Background] Lally P, van Jaarsveld CHM, Potts HWW, Wardle J. How are habits formed: Modelling habit formation in the real world. Eur J Soc Psychology. 2010; 40:998-1009.
- [Background] Litvin S, Saunders R, Maier MA, Luttke S. Gamification as an approach to improve resilience and reduce attrition in mobile mental health interventions: A randomized controlled trial. PLoS One. 2020 Sep 2;15(9):e0237220. doi: 10.1371/journal.pone.0237220. eCollection 2020. PMID 32877425
- [Background] Marin-Gomez FX, Garcia-Moreno Marchan R, Mayos-Fernandez A, Flores-Mateo G, Granado-Font E, Barrera Uriarte ML, Duch J, Rey-Renones C. Exploring Efficacy of a Serious Game (Tobbstop) for Smoking Cessation During Pregnancy: Randomized Controlled Trial. JMIR Serious Games. 2019 Mar 27;7(1):e12835. doi: 10.2196/12835. PMID 30916655
- [Background] Moher D, Shamseer L, Clarke M, Ghersi D, Liberati A, Petticrew M, Shekelle P, Stewart LA; PRISMA-P Group. Preferred reporting items for systematic review and meta-analysis protocols (PRISMA-P) 2015 statement. Syst Rev. 2015 Jan 1;4(1):1. doi: 10.1186/2046-4053-4-1. PMID 25554246
- [Background] Patel MS, Small DS, Harrison JD, Fortunato MP, Oon AL, Rareshide CAL, Reh G, Szwartz G, Guszcza J, Steier D, Kalra P, Hilbert V. Effectiveness of Behaviorally Designed Gamification Interventions With Social Incentives for Increasing Physical Activity Among Overweight and Obese Adults Across the United States: The STEP UP Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1624-1632. doi: 10.1001/jamainternmed.2019.3505. PMID 31498375
- [Background] Statistics Canada. Canadian Internet Use Survey. Last modified: 29 October 2019. Retrieved: 20 October 2020. Available from: https://www150.statcan.gc.ca/n1/dailyquotidien/191029/dq191029a-eng.htm
- [Background] Villinger K, Wahl DR, Boeing H, Schupp HT, Renner B. The effectiveness of app-based mobile interventions on nutrition behaviours and nutrition-related health outcomes: A systematic review and meta-analysis. Obes Rev. 2019 Oct;20(10):1465-1484. doi: 10.1111/obr.12903. Epub 2019 Jul 28. PMID 31353783
- [Derived] Nishi SK, Kavanagh ME, Ramboanga K, Ayoub-Charette S, Modol S, Dias GM, Kendall CWC, Sievenpiper JL, Chiavaroli L. Effect of digital health applications with or without gamification on physical activity and cardiometabolic risk factors: a systematic review and meta-analysis of randomized controlled trials. EClinicalMedicine. 2024 Sep 25;76:102798. doi: 10.1016/j.eclinm.2024.102798. eCollection 2024 Oct. PMID 39764571